CLINICAL TRIAL: NCT05334199
Title: Evaluation of Treatment With Biodegradable Airway Stent for Post Lung Transplant Airway Complication
Brief Title: Biodegradable Airway Stent Post Lung Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: AIDS Malignancy Consortium (Network)
Responsible Party: Principal Investigator, Dirk-Jan Slebos, Prof. dr., University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20220075
Record Dates: First submitted 2022-03-31; First posted 2022-04-19 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Airway Complications Post Lung Transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biodegradable stent treatment group (Experimental): Biodegradable stent treatment group
  Interventions: Device: Biodegradable stent

INTERVENTIONS:
Device: Biodegradable stent — Bronchoscopic placement of biodegradable stent in patients with airway complications after lung transplant

SUMMARY:
Introduction and rationale

Benign airway stenosis or malacia is a frequent complication of lung transplantation occurring in 4-24% of patients, most often occurring two to nine months post-transplant. Initial therapeutic approach consists of conservative endobronchial treatment with recurrent balloon dilatation, radial incision, and electro cautery. For severe case of recurrent stenosis or malacia, airway stent placement can be considered. Different types of airway stent exist, for instance self-extendable metallic stent (SEMS), silicone stent and biodegradable airway stent. Conventional airway stents (SEMS, silicone) are associated with complications as granulation tissue and recurrent infections and can be difficult to remove. Newly developed biodegrabale stents are made of polydioxanone and disintegrate after a period of time are thought to have less side effects, and has been standard of care for the last few years. A sub selection of patients have been treated with conventional stent before treated with biodegradable stent.

Research question

* To assess the efficacy and efficiency of biodegradable airway stent.
* Compare occurrence of adverse events such as infection, dislocation, in stent granulation and difficulty of removal to conventional metallic or silicone stents.
* Asses if biodegradable stent lead to improvement of lung function.
* Assessment of the life span of biodegradable stents.

DETAILED DESCRIPTION:
* Background Recurrent airway stenosis or malacia can be treated with airway stents. Conventional airway stents, for instance self-extendable metallic stent (SEMS) and silicone stent are associated with adverse events as recurrent infection or granulation tissue and can be difficult to remove because of in stent-granulation. Therefore they are used with restraint for benign airway problems. Biodegradable stents are made of polydioxanone and disintegrate after a period of time. They are thought to be well tolerated and associated with less adverse events compared to traditional airway stent and have been used as standard care for multiple years.
* Main research question

  * To assess the efficacy and efficiency of biodegradable airway stent
  * Compare occurrence of adverse events such as infection, dislocation, in stent granulation and difficulty of removal to conventional metallic or silicone stents.
  * Asses if biodegradable stent lead to improvement of lung function.
  * Assessment of the life span of biodegradable stents.
* Design (including population, confounders/outcomes) Retrospective cohort study of patients with airway stenosis or malacia treated with biodegradable airway stent from 2019 in the UMCG and Amsterdam UMC.
* Expected results

  * Less adverse events, hospital admittance and need for bronchoscopic interventions compared to patients treated with conventional stents. No complications associated with removal of stents.
  * Life span around 4 months

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent a lung transplantation and developed airway stenosis or malacia with airway stent requirement

Exclusion Criteria:

* No

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Adverse events | 4 months after placement
  Adverse events associated with airway stents

SECONDARY OUTCOMES:
Change in FEV1 | 1 week post placement
  Change in FEV1 measured by spirometry pre and post stent placement
Change in FVC | 1 week post placement
  Change in FVC measured by spirometry pre and post stent placement
Time to need for new stent placement | 6 months after placement
  Endurance and life span of biodegradable stent measured by time to need for new stent placement

CONTACTS AND LOCATIONS:
Overall Officials: Dirk-Jan Slebos, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (2):
- Netherlands (2):
  - AMC, Amsterdam
  - UMCG, Groningen

IPD SHARING:
Plan to Share IPD: No